CLINICAL TRIAL: NCT05376241
Title: Understanding Affective Processing of Scientific Evidence to Promote Informed Choice for Breast Cancer Screening
Brief Title: Promoting Informed Choice for Breast Cancer Screening
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 20-1866.cc; R37CA254926 (NIH)
Record Dates: First submitted 2022-03-17; First posted 2022-05-17 (Actual); Results first posted 2025-10-24 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Breast Cancer
Keywords: Breast Cancer Screening
MeSH Terms: conditions — Breast Neoplasms | interventions — Decision Support Techniques

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Women age 39-49 in the United States: The group is women age 39-49 in the United States who receive a decision aid intervention. The intervention is a breast cancer screening decision aid with information about screening guidelines, breast cancer mortality reduction, false positives, overdiagnosis, and a personal breast cancer risk estimate.
  Interventions: Behavioral: Decision aid

INTERVENTIONS:
Behavioral: Decision aid — Mammography screening decision aid for women in their 40s with information about screening guidelines, breast cancer mortality reduction, false positives, overdiagnosis, and a personal breast cancer risk estimate.

SUMMARY:
Identify the prevalence and predictors of reactance, self-exemption, disbelief, source derogation in reaction to evidence about mammography benefits and harms, and consequences for decision-making and trust.

DETAILED DESCRIPTION:
In this study, the goal is to identify the prevalence and predictors of reactance, self-exemption, disbelief, and source derogation in reaction to evidence about mammography benefits and harms, and consequences for decision-making and trust. Research has not yet systematically identified the proportion of women who respond negatively (vs. positively) to evidence about the benefits and harms of mammography screening, or attempted to explain these responses by examining theory-driven predictors. The Investigator will develop and conduct a probability-based nationally representative survey in which mammography evidence is communicated using current best practices in risk communication. The Investigators will identify theory-driven predictors of negative and positive responses to that evidence, and identify consequences of these responses for screening decision-making and trust.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Between 39-49 years of age
* No history of breast cancer
* No known BRCA 1/2 mutation

Exclusion Criteria:

* Non-English or Spanish Speaking
* Persons unable to provide informed consent (e.g. sever dementia or cognitive disability or illiterate
* History of breast cancer
* Known BRCA 1/2 mutation

Ages: 39 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Female
Study Population: Women age 39-49 in the United States.
Sampling Method: Probability Sample
Enrollment: 637 (Actual)
Dates: Start 2020-08-07 (Actual); Primary Completion 2023-05-07 (Actual); Study Completion 2023-05-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laura Scherer, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Anschutz Medical Campus, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified survey data will be shared using the Open Science Framework. These data will be shared with reviewers and editors prior to publication of main results. After publication of main results, deidentified data will be made available publicly.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: All elements of the study except data will be shared immediately. Survey data will be shared with reviewers and editors prior to publication of main study results. Survey data will be shared publicly after publication of main study results.
URL: https://osf.io/y8stc/

REFERENCES:
- [Background] Scherer LD, Lewis CL, Cappella JN, Hersch J, McCaffery K, Tate C, Smyth HL, Mosley B, Morse B, Schapira MM. Skeptical reactions to breast cancer screening benefits and harms: Antecedents, consequences, and implications for screening communication. Health Psychol. 2025 Jun;44(6):608-619. doi: 10.1037/hea0001442. Epub 2024 Nov 25. PMID 39585772
- [Background] Scherer LD, Lewis CL, McCaffery K, Hersch J, Cappella JN, Tate C, Morse B, Arnett K, Mosley B, Smyth HL, Schapira MM. Mammography Screening Preferences Among Screening-Eligible Women in Their 40s : A National U.S. Survey. Ann Intern Med. 2024 Aug;177(8):1069-1077. doi: 10.7326/M23-3325. Epub 2024 Jul 16. PMID 39008858
- [Background] Parmet T, Yoder G, Morse B, Cappella J, Schapira M, Lewis C, McCaffery K, Smyth H, Hersch J, Scherer LD. Trust in the healthcare system declines after exposure to information about the harms and benefits of breast cancer screening. J Health Psychol. 2025 Nov;30(13):4091-4097. doi: 10.1177/13591053251315383. Epub 2025 Feb 7. PMID 39917819
- [Result] Morse B, Parmet T, Yoder G, Tate CE, Lewis CL, McCaffery K, Cappella JN, Hersch J, Schapira MM, Scherer LD. Evaluation of how US women react to a decision aid informing them of the harms and benefits of mammography: a qualitative study. BMJ Open. 2025 Mar 18;15(3):e087997. doi: 10.1136/bmjopen-2024-087997. PMID 40107692
- Available data/document: Individual Participant Data Set — https://osf.io/y8stc/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Data were collected from January to April 2022 through the online survey research panel Ipsos KnowledgePanel. A total of 637 participants were identified for the survey, but 22 did not meet eligibility criteria, 103 did not complete the survey, and 17 were excluded for failing 2 attention check questions, resulting in a final analytic sample of 495 participants.
Period: Overall Study
Arm/Group | Women Age 39-49 in the United States
Started | 637
Completed | 495
Not Completed | 142
Not completed — did not meet eligibility criteria after consenting | 22
Not completed — 103 did not complete the survey | 103
Not completed — 17 failed 2 attention check questions | 17

BASELINE CHARACTERISTICS:
Population: Analytic sample was N=495, due to 17 participants excluded for failing 2 attention check questions
Arm/Group | Women Age 39-49 in the United States
Number analyzed (Participants) | 495
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.9 (3.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 495
  Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Non-hispanic white | 327
  non-hispanic Black | 53
  non-hispanic other race | 25
  non-hispanic >2 races | 20
  Hispanic | 70

OUTCOME MEASURES:

1. Primary Outcome: Reactance
Description: In response to mammography evidence, feeling that the information is manipulative or biased. 4 questions total, each on a 7 point Likert scale, with mean scores that range from 1 to 5. Higher mean scores reflect greater reactance.
Time Frame: 24 hours
Population: The group is women aged 39-49 in the United States with no history of breast cancer or known BRCA1/2 mutation, who receive a decision aid intervention. The intervention is a breast cancer screening decision aid with information about screening guidelines, breast cancer mortality reduction, false positives, overdiagnosis, and a personal breast cancer risk estimate.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Women Age 39-49 in the United States
Number analyzed (Participants) | 495
score on a scale
  Response to screening benefits | 2.28 (0.71)
  Response to false positives | 2.45 (0.75)
  Response to overdiagnosis | 2.55 (0.80)

2. Primary Outcome: Disbelief
Description: In response to mammography evidence, feeling that the evidence is not accurate or believable. 4 questions total, each on a 5 point Likert scale, with mean scores that range from 1 to 5. Higher mean score reflects more disbelief in the information.
Time Frame: 24 hours
Population: The group is women age 39-49 in the United States who receive a decision aid intervention. The intervention is a breast cancer screening decision aid with information about screening guidelines, breast cancer mortality reduction, false positives, overdiagnosis, and a personal breast cancer risk estimate.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Women Age 39-49 in the United States
Number analyzed (Participants) | 495
Score on a scale
  Response to screening benefits | 2.06 (0.61)
  Response to false positives | 2.32 (0.63)
  Response to overdiagnosis | 2.41 (0.68)

3. Primary Outcome: Source Derogation
Description: In response to mammography evidence, feeling that the source of the evidence is not trustworthy or competent. 4 questions total, each on a 5 point Likert scale, with mean scores that range from 1 to 5. Higher mean score reflects more source derogation.
Time Frame: 24 hours
Population: as for outcome 2
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Women Age 39-49 in the United States
Number analyzed (Participants) | 495
score on a scale | 2.56 (0.09)

4. Primary Outcome: Self Exemption
Description: Feeling that mammography evidence is not relevant to oneself.34 questions total, each on a 5 point Likert scale, with mean scores that range from 1 to 5. Higher mean scores indicate greater belief that the information is not self relevant.
Time Frame: 24 hours
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Women Age 39-49 in the United States
Number analyzed (Participants) | 495
score on a scale
  Response to screening benefits | 2.20 (0.70)
  Response to false positives | 2.21 (0.71)
  Response to overdiagnosis | 2.32 (0.72)

5. Primary Outcome: Screening Intentions
Description: Intentions to engage in mammography screening. Options will include: 1. I am planning to start/continue having regular mammograms this year. 2. I am planning to wait until I'm older but before age 50 to have my first/next mammogram. 3. I am planning to wait until I am 50 to have my first/next mammogram. 4. I am not planning to have a mammogram in the future at any age
Time Frame: 24 hours
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Women Age 39-49 in the United States
Number analyzed (Participants) | 495
Participants
  Have regular mammograms at current age | 286
  Wait until older but before age 50 | 100
  Wait until age 50 | 88
  never have a mammogram | 21

6. Secondary Outcome: Medical Mistrust Scale (Eaton et al., 2015)
Description: 6 question scale that assesses mistrust in healthcare providers. Calculated as mean trust (range 1-low trust to 5-high trust). Assessed both pre and post receipt of screening decision aid to evaluate change
Time Frame: 24 hours
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Women Age 39-49 in the United States
Number analyzed (Participants) | 495
score on a scale
  Pre-DA trust | 3.11 (0.69)
  Post-DA trust | 3.02 (0.65)

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Women Age 39-49 in the United States
All-Cause Mortality (participants affected / at risk) | 0/495
Serious Adverse Events (participants affected / at risk) | 0/495
Other Adverse Events (participants affected / at risk) | 0/495

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-05-10): https://cdn.clinicaltrials.gov/large-docs/41/NCT05376241/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-10): https://cdn.clinicaltrials.gov/large-docs/41/NCT05376241/SAP_001.pdf